CLINICAL TRIAL: NCT01079962
Title: A Prospective, Multi-center, Randomized, Open-label, Clinical Trial to Compare the Aortic Pulse Pressure Effects of Bisoprolol and Atenolol in 12 Weeks Treatment of Hypertension
Brief Title: An Active-controlled, Clinical Trial to Assess Central Hemodynamic Effects of Bisoprolol in Hypertensive Patients (Central Hemodynamic Assessment Measured in Patient With HypertensION [CHAMPION])
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD 084000-505
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2012-10-02 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Bisoprolol; Atenolol; Hypertension; Blood pressure
MeSH Terms: conditions — Hypertension | interventions — Bisoprolol; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bisoprolol (Experimental)
  Interventions: Drug: Bisoprolol
- Atenolol (Active Comparator)
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Bisoprolol — Bisoprolol tablet will be administered orally at a dose of 5 milligram (mg) once daily in the morning for 12 weeks.
  Other Names: CONCOR®
  Arms: Bisoprolol
Drug: Atenolol — Atenolol tablet will be administered orally at a dose of 50 mg once daily in the morning for 12 weeks.
  Other Names: TENORMIN®
  Arms: Atenolol

SUMMARY:
Antihypertensive drugs aim to reduce blood pressure (BP) either through decrease of the total peripheral resistance through vasodilatation at the level of arterioles (microcirculation) or by decreasing the cardiac output through reduction of the stroke volume or heart rate or both. On the other hand, all antihypertensive drugs might potentially decrease arterial stiffness passively with the reduction of the distending pressure or with the resynchronization of the reflected pressure wave. With theses potential mechanisms, it is also expected that these drugs might exert a favorable effect on pulse pressure amplification between central and peripheral arteries.

However, there is solid evidence that the widely applied antihypertensive drugs have differential effect on brachial and central BP. Several reports in the past have confirmed the potential hypothesis that beta blockers decrease central BP less than the observed reduction at the level of the brachial artery. It has been hypothesized that deceleration of heart rate and the re synchronizing the reflected pressure wave earlier in the systolic phase seems to be the leading cause of non-favorable effect of beta blockers on central BP, these effects might be partially counterbalanced in beta blockers with high beta-1 selectivity resulting in less peripheral vasoconstriction properties.

DETAILED DESCRIPTION:
Central pulse pressure is a better predictor of left ventricular mass and carotid intima thickness, and the conventional peripheral BP does not seem to be an accurate reflection of central arterial BP. The pulse pressure amplification between peripheral and central arteries reflects the left ventricular afterload, subendothelial viability, and the intensity of cyclic stress imposed to the renal and cerebral micro- and macro vessels. As central hemodynamic parameters are independently associated with organ damage and are closely related to important cardiovascular outcome, it is suggested that the new clinical trials on antihypertensive drug treatment should compare simultaneously the chronic effect of drugs on both peripheral and central BP.

OBJECTIVES

Primary objective:

* To assess the effect of bisoprolol versus atenolol on the aortic pulse pressure as a central hemodynamic index in subjects with hypertension

Secondary objectives:

* To assess the effect of bisoprolol versus atenolol on the aortic BP as a central hemodynamic index in subjects with hypertension
* To assess the effect of bisoprolol versus atenolol on the AIx and cfPWV as arterial stiffness indexes in subjects with hypertension
* To assess the effect of bisoprolol versus atenolol on the aortic pulse pressure as a central hemodynamic index at interim visit (Visit 4)
* To assess the effect of bisoprolol versus atenolol on the lipid profile and serum glucose as metabolism indexes
* To assess the effect of bisoprolol versus atenolol on the brachial BP as a peripheral BP index in subjects with hypertension
* To assess the safety and tolerability of bisoprolol versus atenolol in subjects with hypertension

The present study will be approximately of 14 weeks duration comprising of 1 week screening, followed by a 12 weeks treatment period and a 2 weeks post study follow up contact conducted via telephone to monitor additional serious adverse experiences.

There will be 4 scheduled visits (at Day -7, Day 0, Week 4 and Week 12). After screening period in which eligibility criteria were confirmed, subjects with hypertension will be randomized in a 1:1 ratio to receive treatment with either bisoprolol or atenolol. Hemodynamic measurements will be made at baseline, Week 4, Week 12 and biochemical measurements will be made at baseline (Day 0) and at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* An antihypertensive-naive subject or a subject who has not been taking the previously administered antihypertensive agent for at least 4 weeks prior to screening
* Subjects aged between 20 and 75 years, inclusive
* Subjects with systolic blood pressure (SBP) greater than or equal to 140 millimeter of mercury (mmHg) and less than 180 mmHg or diastolic blood pressure (DBP) greater than or equal to 90 mmHg and less than 110 mmHg

Exclusion Criteria:

* Subjects with secondary hypertension
* Subjects with renal impairment (Creatinine greater than 150 micromoles/liter [mcmol/L] or Creatinine greater than 1.7 mg/deciliter [dL])
* Subjects with severe hypertension (Stage III) SBP greater than or equal to 180 mmHg or DBP greater than or equal to 110 mmHg
* Subjects with congestive heart failure, acute myocardial infarction, unstable angina
* Subjects with moderate bronchial asthma, chronic obstructive pulmonary disease
* Subjects with symptomatic bradycardia, radial artery injury, second degree or third degree atrioventricular (AV) block, atrial fibrillation, atrial flutter, left bundle branch block (LBBB)
* Subjects with a history of hypersensitivity to bisoprolol and atenolol products
* Pregnancy or breastfeeding women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Ltd., Korea, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Severance Hosptial, 250, Seongsanno, Seodaemungu, Seoul, South Korea

REFERENCES:
- [Derived] Park S, Rhee MY, Lee SY, Park SW, Jeon D, Kim BW, Kwan J, Choi D. A prospective, randomized, open-label, active-controlled, clinical trial to assess central haemodynamic effects of bisoprolol and atenolol in hypertensive patients. J Hypertens. 2013 Apr;31(4):813-9. doi: 10.1097/HJH.0b013e32835e8f5b. PMID 23385648

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 228 participants were screened for the study, out of which 19 were screen failures and 209 participants received the study medication.
Groups:
- Bisoprolol: Single dose of bisoprolol tablet (CONCOR®) administered orally at a dose of 5 milligram (mg) daily every morning for 12 weeks.
- Atenolol: Single dose of atenolol tablet (TENORMIN®) administered orally at a dose of 50 mg daily every morning for 12 weeks.
Period: Overall Study
Arm/Group | Bisoprolol | Atenolol
Started | 105 | 104
Completed | 90 | 89
Not Completed | 15 | 15
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Protocol Violation | 2 | 2
Not completed — No blood pressure (BP) control | 3 | 0
Not completed — Inclusion/exclusion criteria | 1 | 3
Not completed — Participant not returning for next visit | 1 | 0
Not completed — Due to arrhythmia/bradycardia | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bisoprolol | Atenolol | Total
Number analyzed (Participants) | 105 | 104 | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (11.2) [25 to 74] | 52.2 (9.3) [21 to 75] | 52.2 (10.2) [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 46 | 85
  Male | 66 | 58 | 124

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Aortic Pulse Pressure (APP) in Intention to Treat (ITT) Population at Week 12
Description: The APP was calculated as aortic systolic pressure minus aortic diastolic pressure. The change in APP at Week 12 was calculated as APP at Week 12 minus APP at baseline.
Time Frame: Baseline and Week 12
Population: ITT population included all participants who had received at least 1 dose of the study medication or comparator and at least 1 post-dose measurement of aortic pulse pressure. "n" signifies those participants who were evaluated for this measure at the specified time point.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 96 | 95
Millimeter of mercury (mmHg)
  Baseline (n=96, 95) | 47.49 (11.33) | 45.93 (11.62)
  Change in APP at Week 12 (n=90, 89) | -4.40 (9.29) | -3.69 (8.86)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Change in APP at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.5943, t-test, 2 sided — No adjustment of p-value was done and priori threshold was 0.05; Mean Difference (Final Values) = 0.701, 95% CI 2-sided [-1.89 to 3.29]

2. Secondary Outcome: Change From Baseline in Aortic Blood Pressure (BP) at Week 4 and Week 12
Description: The change in aortic BP (aortic systolic blood pressure [SBP], aortic diastolic blood pressure [DBP] and aortic mean blood pressure [BP]) at Week 4 and Week 12 was calculated as aortic BP (aortic SBP, aortic DBP and aortic mean BP) at Week 4 and Week 12 minus aortic BP (aortic SBP, aortic DBP and aortic mean BP) at baseline.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 96 | 95
mmHg
  Change in aortic SBP at Week 4 (n=96, 95) | -13.90 (12.68) | -13.57 (12.73)
  Change in aortic SBP at Week 12 (n=90, 89) | -15.34 (15.11) | -12.71 (14.67)
  Change in aortic DBP at Week 4 (n=96, 95) | -10.86 (8.23) | -9.47 (8.23)
  Change in aortic DBP at Week 12 (n=90, 89) | -10.94 (9.53) | -9.01 (8.79)
  Change in aortic mean BP at Week 4 (n=96, 95) | -11.88 (8.60) | -10.84 (9.07)
  Change in aortic mean BP at Week 12 (n=90, 89) | -12.41 (10.84) | -10.24 (10.28)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Change in SBP at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.8589, t-test, 2 sided
Statistical Analysis 2: Comparison: Bisoprolol vs Atenolol; Change in SBP at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.2223, t-test, 2 sided
Statistical Analysis 3: Comparison: Bisoprolol vs Atenolol; Change in DBP at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.2443, t-test, 2 sided
Statistical Analysis 4: Comparison: Bisoprolol vs Atenolol; Change in DBP at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.1481, t-test, 2 sided
Statistical Analysis 5: Comparison: Bisoprolol vs Atenolol; Change in mean BP at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.4188, t-test, 2 sided
Statistical Analysis 6: Comparison: Bisoprolol vs Atenolol; Change in mean BP at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.1586, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Aortic Augmentation Index (AIx) at Week 4 and Week 12
Description: Augmentation index is a composite measure of wave reflection and systemic arterial stiffness which was calculated as the difference between the second and first systolic peaks. The change in AIx at Week 4 and Week 12 was calculated as AIx at Week 4 and Week 12 minus AIx at baseline.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 96 | 95
Ratio
  Change in AIx at Week 4 (n=96, 95) | -1.56 (10.43) | -0.01 (10.14)
  Change in AIx at Week 12 (n=90, 89) | 0.61 (9.18) | 1.21 (9.41)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Change in AIx at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.2987, t-test, 2 sided
Statistical Analysis 2: Comparison: Bisoprolol vs Atenolol; Change in AIx at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.6584, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Carotid-femoral Pulse Wave Velocity (cfPWV) at Week 4 and Week 12
Description: Pulse wave velocity (PWV) is used as a measure of arterial stiffness, which is a measure of the cushioning functioning of major vessels like the aorta. The velocity of the Pulse wave (PW) along an artery is dependent on the stiffness of that artery. The change in cfPWV at Week 4 and Week 12 was calculated as cfPWV at Week 4 and Week 12 minus cfPWV at baseline.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters per second (m/s)
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 96 | 95
Meters per second (m/s)
  Change in cfPWV at Week 4 (n=96, 95) | -0.60 (1.33) | -0.81 (1.15)
  Change cfPWV at Week 12 (n=90, 89) | -0.72 (1.40) | -0.87 (1.56)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Change in cfPWV at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.2511, t-test, 2 sided
Statistical Analysis 2: Comparison: Bisoprolol vs Atenolol; Change in cfPWV at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.5007, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Heart Rate at Week 4 and Week 12
Description: The change in heart rate at Week 4 and Week 12 was calculated as heart rate at Week 4 and Week 12 minus heart rate at baseline.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 96 | 95
Beats per minute (bpm)
  Change in heart rate at Week 4 (n= 96, 95) | -6.21 (7.72) | -6.20 (8.25)
  Change heart rate at Week 12 (n= 90, 89) | -8.64 (7.95) | -7.84 (9.15)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Change in heart rate at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.9943, t-test, 2 sided
Statistical Analysis 2: Comparison: Bisoprolol vs Atenolol; Change in heart rate at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.5230, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in Aortic Pulse Pressure (APP) at Week 4
Description: The APP was calculated as aortic systolic pressure minus aortic diastolic pressure. The change in APP at Week 4 was calculated as APP at Week 4 minus APP at baseline.
Time Frame: Baseline and Week 4
Population: ITT population included all participants who had received at least 1 dose of the study medication or comparator and at least 1 post-dose measurement of aortic pulse pressure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 96 | 95
mmHg | -3.02 (10.56) | -4.09 (8.72)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Test type: Superiority or Other; p = 0.4447, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Lipid Levels at Week 12
Description: The lipid levels evaluated were total cholesterol, low density lipoprotein (LDL) cholesterol, and high density lipoprotein (HDL) cholesterol blood concentrations. The change in lipid levels at Week 12 was calculated as lipid levels at Week 12 minus lipid levels at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milligram/decilitre (mg/dL)
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 96 | 95
Milligram/decilitre (mg/dL)
  Change in Total cholesterol at Week 12 | -3.43 (23.35) | -0.37 (24.79)
  Change in LDL-cholesterol at Week 12 | -2.29 (19.01) | 1.31 (17.77)
  Change in HDL-cholesterol at Week 12 | -1.58 (7.13) | -3.02 (7.54)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Change in Total cholesterol at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.3960, t-test, 2 sided
Statistical Analysis 2: Comparison: Bisoprolol vs Atenolol; Change in LDL-cholesterol at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.1919, t-test, 2 sided
Statistical Analysis 3: Comparison: Bisoprolol vs Atenolol; Change in HDL-cholesterol at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.1896, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Blood Glucose Levels at Week 12
Description: The change in blood glucose level at Week 12 was calculated as blood glucose level at Week 12 minus blood glucose level at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 90 | 89
Millimoles per liter (mmol/L) | -0.23 (17.85) | -0.45 (12.03)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Test type: Superiority or Other; p = 0.9244, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Brachial Blood Pressure (BP) at Week 4 and Week 12
Description: The change in brachial BP (brachial SBP, brachial DBP and brachial mean BP) at Week 4 and Week 12 was calculated as brachial BP (brachial SBP, brachial DBP and brachial mean BP) at Week 4 and Week 12 minus brachial BP (brachial SBP, brachial DBP and brachial mean BP) at baseline.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 96 | 95
mmHg
  Change in brachial SBP at Week 4 (n=96, 95) | -17.45 (11.74) | -17.52 (12.53)
  Change in brachial SBP at Week 12 (n=90, 89) | -19.10 (14.55) | -17.63 (13.74)
  Change in brachial DBP at Week 4 (n=96, 95) | -12.70 (9.01) | -11.36 (8.34)
  Change in brachial DBP at Week 12 (n=90, 89) | -13.39 (9.90) | -10.61 (8.79)
  Change in brachial mean BP at Week 4 (n=96, 95) | -14.28 (9.28) | -13.41 (8.94)
  Change in brachial mean BP at Week 12 (n=90, 89) | -15.29 (10.78) | -12.95 (9.96)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Change in SBP at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.9692, t-test, 2 sided
Statistical Analysis 2: Comparison: Bisoprolol vs Atenolol; Change in SBP at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.4731, t-test, 2 sided
Statistical Analysis 3: Comparison: Bisoprolol vs Atenolol; Change in DBP at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.2876, t-test, 2 sided
Statistical Analysis 4: Comparison: Bisoprolol vs Atenolol; Change in DBP at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.0420, t-test, 2 sided
Statistical Analysis 5: Comparison: Bisoprolol vs Atenolol; Change in mean BP at Week 4: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.5100, t-test, 2 sided
Statistical Analysis 6: Comparison: Bisoprolol vs Atenolol; Change in mean BP at Week 12: p-value was calculated by 2 sided t-test; Test type: Superiority or Other; p = 0.1207, t-test, 2 sided

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Time Frame: Baseline up to Week 14 (follow-up visit)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 105 | 104
Participants | 36 | 32

11. Primary Outcome: Change From Baseline in Aortic Pulse Pressure (APP) in Per Protocol (PP) Population at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Per protocol (PP) population included those participants for whom primary and secondary efficacy endpoints were all measured, and who did not meet the withdrawal criteria and showed 75 percent of medication compliance.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol | Atenolol
Number analyzed (Participants) | 85 | 89
mmHg
  Baseline | 46.87 (11.34) | 46.53 (11.66)
  Change in APP at Week 12 | -4.33 (9.66) | -3.89 (9.07)
Statistical Analysis 1: Comparison: Bisoprolol vs Atenolol; Test type: Superiority or Other; p = 0.7561, t-test, 2 sided — No adjustment of p-value was done and priori threshold was 0.05; Mean Difference (Final Values) = 0.442, 95% CI [-2.36 to 3.24]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 14 (follow-up visit)
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Bisoprolol | Atenolol
Serious Adverse Events (participants affected / at risk) | 7/105 | 3/104
Other Adverse Events (participants affected / at risk) | 29/105 | 29/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=105) | Atenolol (N=104)
Concussion (General disorders) | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Tendon rupture (Musculoskeletal and connective tissue disorders) | 1 | 0
Uterine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Coronary artery disorder (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Headache aggravated (Nervous system disorders) | 1 | 0
Dizziness aggravated (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=105) | Atenolol (N=104)
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1
Liver fatty (Hepatobiliary disorders) | 0 | 2
Cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia aggravated (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain neck/shoulder (Musculoskeletal and connective tissue disorders) | 1 | 0
Cartilage damage (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain aggravated (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperlipaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Common cold (General disorders) | 2 | 6
Bronchitis (General disorders) | 0 | 1
Herpes zoster (General disorders) | 0 | 1
Cystitis (General disorders) | 1 | 0
Tinea (General disorders) | 1 | 0
Upper respiratory tract infection (General disorders) | 1 | 2
Otitis media (General disorders) | 1 | 0
Impotence (Reproductive system and breast disorders) | 0 | 1
Dry eyes (Eye disorders) | 0 | 1
Uterine fibromyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
AV block first degree (General disorders) | 1 | 0
Sinus bradycardia (General disorders) | 3 | 4
Bradyarrhythmia (General disorders) | 2 | 1
Cardiomegaly (Cardiac disorders) | 1 | 0
Bladder irritability (General disorders) | 1 | 0
Ureteral calculus (General disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Polyposis gastric (Gastrointestinal disorders) | 1 | 0
Anaemia (General disorders) | 2 | 0
Chest tightness of (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 2
Chest pressure sensation of (General disorders) | 0 | 1
Chest pain (General disorders) | 4 | 0
Oedema (General disorders) | 1 | 0
Pain groin (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Hot flushes (General disorders) | 0 | 1
Pain in limb (General disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 2
Sleepiness (Psychiatric disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Eyelid fluttering (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Headache aggravated (Nervous system disorders) | 1 | 0
Radiculopathy cervical (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 8 | 6
Itching (Skin and subcutaneous tissue disorders) | 2 | 0
Sweating increased (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin cysts (Skin and subcutaneous tissue disorders) | 1 | 0
Rhinitis allergic atopic (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other